CLINICAL TRIAL: NCT00380302
Title: A Double-Blind Placebo-Controlled Study of the Activity of AVE1625 at Doses of 10 mg and 40mg for 12 Weeks in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Activity of AVE1625 in Mild to Moderate Alzheimer's Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT10019; EUDRACT: 2006-002317-12
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; symptomatic; cognition
MeSH Terms: conditions — Alzheimer Disease | interventions — AVE1625

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: AVE1625

SUMMARY:
Primary: This study is being conducted to evaluate if AVE1625 is safe and tolerated in patients with Alzheimer's disease that is not too severe. There is also evaluation of whether patients who take the study medication improve compared to patients who take a placebo (sugar pill).

Secondary:The study will also evaluate the blood levels of the study medication, AVE1625 in patients who join the study.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of Alzheimer's disease
* Recent brain image(Computerized Axial Tomographic Scan -CAT scan or Magnetic Resonance Imaging - MRI)
* Mild to moderate range of disease; not too severe

Exclusion Criteria:

* Severe or unstable medical diseases
* Neurological disorder other than Alzheimer's disease
* Depression that is not well controlled
* Treatment with memantine
* Inpatient in a total care facility (e.g.: Nursing home)
* Lack of reliable caregiver

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability throughout the study:adverse events collected by spontaneous report
physical examination and neurological assessment
vital sign monitoring, clinical laboratories, and ECGs.
Efficacy variables:measures of change in cognition, global functioning and behavior at week 12.

SECONDARY OUTCOMES:
Pharmacokinetic parameters will be assessed throughout the 12-week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Bromma, Sweden

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com